CLINICAL TRIAL: NCT06308003
Title: Effect of Surgical Approach on Postoperative Bleeding in Patients Undergoing Hip Arthroplasty: Anterior Vs. Posterolateral Route
Brief Title: Effect of Surgical Approach on Postoperative Bleeding in Patien Arthroplasty
Status: Recruiting | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: PTA CONF
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Hip Arthropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Anterior hip arthroplasty — Anterior hip arthroplasty

SUMMARY:
The study is, in accordance with current legislation, definable as monocentric Prospective Observational.

The primary outcome will be blood loss calculated on the basis of hemoglobin (Hb) on the third postoperative day.

adult patients who will undergo surgery of hip arthroplasty.

Patients will undergo:

Preoperative T0: clinical visit/medical history, completion of the VAS questionnaire, Blood sampling to assess hemoglobin values Operative T1: hip arthroplasty surgery using one of the surgical approaches routinely used within our Institute T2 - Postoperative at 1 day from T1: VAS questionnaire, evaluation of any Adverse events T3 - Postoperative at 3 days from T1: blood loss based on the values of hemoglobin (Hb), assessment of any adverse events, and VAS questionnaire T4- Post operative at 45 days +/- 10 days from T1: evaluation of any events adverse, follow-up visit.

DETAILED DESCRIPTION:
The presence of bleeding and pain after prosthesis surgery Hip injuries can affect the patient's condition in the postoperative period increasing the length of hospital stay and slowing down the rehabilitation process.

It is hypothesized that there are differences in terms of postoperative bleeding, Postoperative pain and hospital stay time between different approaches surgical procedures in the treatment of hip osteoarthritis with arthroprosthesis. The adoption of a Surgical approach that can reduce bleeding and pain could reduce the length of hospital stay in patients undergoing hip arthroplasty.

The primary outcome will be blood loss calculated on the basis of hemoglobin (Hb) on the third postoperative day.

Secondary objectives are postoperative pain assessment with questionnaire VAS and length of hospital stay according to surgical approach used (anterior Vs. posterolateral route). Also evaluate Any adverse events.

Adult patients who will undergo surgery of hip arthroplasty.

The inclusion criteria are:

* adult patients with coxarthrosis who are candidates for surgery hip arthroplasty
* Signing of the Informed Consent and consent to collaborate in all study procedures.

The exclusion criteria are:

* Minors
* Pregnant women (self-declaration)
* patients with BMI ≥ 30
* Non-acceptance of informed consent
* Patients with prior unilateral hip reconstructive surgery or Contralateral

ELIGIBILITY:
Inclusion Criteria:

* adult patients with coxarthrosis who are candidates for surgery hip arthroplasty
* Signing of the Informed Consent and consent to collaborate in all study procedures.

Exclusion Criteria:

* Minors
* Pregnant women (self-declaration)
* patients with BMI ≥ 30
* Non-acceptance of informed consent
* Patients with prior unilateral hip reconstructive surgery or Contralateral

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients who will undergo surgery of hip arthroplasty
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will be blood loss calculated on the basis of hemoglobin (Hb) on the third postoperative day. | the third postoperative day
  The primary outcome will be blood loss calculated on the basis of hemoglobin (Hb) on the third postoperative day.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Ventura, Principal Investigator — Ospedale Galeazzi-Sant'Ambrogio
Locations (1):
- Istituto Clinico San Siro, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided